CLINICAL TRIAL: NCT00616642
Title: Rosiglitazone (Peroxisome Proliferating Activating Receptor-gamma {PPAR-y} Ligand) Treatment of Pituitary Tumors
Brief Title: Rosiglitazone in Treating Patients With Pituitary Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low patient recruitment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000586480; UCLA-0411082-03
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Results first posted 2013-04-15 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2013-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent pituitary tumor; ACTH-producing pituitary tumor; nonfunctioning pituitary tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Pituitary Neoplasms | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (ACTH-secreting adenomas) (Experimental): Patients receive 4 mg oral rosiglitazone maleate once daily in week 1 and then 8 mg once daily beginning in week 2 and continuing for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: rosiglitazone maleate
- Group 2 (non-secreting macroadenomas) (Experimental): Patients receive 4 mg oral rosiglitazone maleate once daily in week 1 and then 8 mg once daily beginning in week 2 and continuing for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: rosiglitazone maleate

INTERVENTIONS:
Drug: rosiglitazone maleate — Given orally

SUMMARY:
RATIONALE: Rosiglitazone may help pituitary adenoma cells become more like normal cells, and grow and spread more slowly.

PURPOSE: This phase II trial is studying how well rosiglitazone works in treating patients with newly diagnosed or residual or recurrent pituitary adenoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the effect of rosiglitazone maleate on the core biochemical parameter, 24-hour urinary free cortisol levels, in patients with recurrent or uncured pituitary-dependent Cushing disease. (Group 1)
* To assess the effect of this drug on corticotropin-releasing hormone-stimulated pituitary tumor ACTH secretion in patients with recurrent or uncured pituitary-dependent Cushing disease. (Group 1)
* To assess the effect of this drug on tumor growth in patients with non-secreting pituitary macroadenoma (> 10 mm) using RECIST criteria. (Group 2)
* To assess the effect of this drug on pituitary tumor gonadotropin (i.e., follicle-stimulating hormone, leuteinizing hormone, and alpha-subunit) secretion in patients with non-secreting macroadenoma. (Group 2)
* To assess the overall safety and tolerability of this drug in both cohorts of patients.
* To assess the overall quality of life, in terms of performance status during treatment, of both cohorts of patients using the Karnofsky performance index.

OUTLINE: Patients are grouped according to adrenocorticotropic hormone (ACTH)-secreting status (yes [Group 1] vs no [Group 2]).

* Group 1 (ACTH-secreting adenomas): Patients receive 4 mg oral rosiglitazone maleate once daily in week 1 and then 8 mg once daily beginning in week 2 and continuing for up to 6 months in the absence of disease progression or unacceptable toxicity.
* Group 2 (non-secreting macroadenomas): Patients receive 4 mg oral rosiglitazone maleate once daily in week 1 and then 8 mg once daily beginning in week 2 and continuing for up to 12 months in the absence of disease progression or unacceptable toxicity.

Patients undergo collection of blood and urine samples at baseline and after completion of study therapy to assess pituitary function, thyroid function, and 24-hour urinary free cortisol levels. Additional assessments include corticotrophin-stimulation testing, dynamic pituitary function testing (i.e., arginine/growth-hormone releasing-hormone testing) to measure growth hormone secretion, and overnight 1 mg dexamethasone suppression testing to measure 8 a.m. serum cortisol levels. Patients also undergo MRI at baseline and after completion of study therapy to examine the effects of rosiglitazone maleate treatment on pituitary tumor size.

Patients complete a questionnaire at baseline and monthly during study for evaluation of headaches.

PROJECTED ACCRUAL: A total of 15 patients with ACTH-secreting pituitary tumor and 15 patients with non-secreting pituitary macroadenomas will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically demonstrable pituitary tumor, including either of the following subtypes:
* ACTH-secreting adenoma
* Residual or recurrent disease ≥ 1 month after prior pituitary surgery

  * Clinically demonstrable tumor, as evidenced by both of the following:

    * Elevated 24-hour urinary free cortisol (UFC) level
    * Lack of suppression of 8 a.m. serum cortisol to < 1.8 µg/dL after administration of dexamethasone 1 mg at 11 p.m. the previous night
  * Tumor demonstrated by MRI performed with and without contrast and/or by inferior petrosal sinus sampling with evidence of a central ACTH source.
* Normal visual field evaluation by Goldman perimetry
* Hypopituitarism allowed as evidenced by any or all of the following:
* Subnormal growth hormone (GH) response to arginine/GH-releasing hormone testing (normal response is an increase of 2-6 ng/me)
* Low age and sex-matched IGF-1 levels
* Low thyroid-stimulating hormone, free triiodothyronine, and free thyroxine levels
* Low estradiol levels
* Low leuteinizing hormone (LH) and low follicle-stimulating hormone (FSH) levels in post-menopausal female patients OR low testosterone, LH, and FSH levels in male patients
* Patients with Cushing disease (i.e., harboring ACTH-secreting pituitary adenomas) must meet the following criteria:
* Hypercortisolemic (i.e., uncured) despite ≥ 1 pituitary surgery
* Refuse to undergo pituitary irradiation and/or bilateral adrenalectomy
* Refuse alternate steroid-lowering therapy such as ketoconazole and/or metyrapone.
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 2 months prior to, during, and for 1 month after completion of study therapy.
* Non-secreting pituitary adenoma

  * Newly diagnosed disease or residual tumor after prior surgical debulking

    * Patients underwent prior surgical debulking must be ≥ 3 months post-surgery
  * More than 10 mm in widest diameter (i.e., macroadenoma), as demonstrated by pituitary MRI performed with and without gadolinium
* Must be able to undergo pituitary MRI (group 2)
* More than 2 months since prior blood donation > 400 mL
* More than 1 month since prior unlicensed drugs or participation in a clinical trial using an investigational drug
* More than 3 months since prior rosiglitazone maleate or other thiazolidinedione
* Patients diagnosed with hypopituitarism (except post-menopausal females) are required to initiate hormone-replacement therapy (HRT) for the 6-month duration of the study and to discontinue HRT at the end of 6 months to re-evaluate hypopituitarism

Exclusion Criteria:

* Acromegaly as demonstrated by normal serum insulin-like growth factor-1 (IGF-1) level
* Cushing disease as demonstrated by normal 24-hour UFC cortisol level
* Prolactinoma as demonstrated by normal to moderately elevated prolactin levels (moderate elevations in serum prolactin [< 200 ng/mL] can occur in non-secreting tumors due to pituitary stalk displacement)

  * clinically significant renal, hematologic, cardiac, or hepatic abnormalities within the past month
  * other active malignancy within the past five years except basal cell carcinoma or carcinoma in situ of the cervix
  * evidence of drug or alcohol abuse
  * prior or current medical condition that may interfere with the conduct of the study or evaluation of its results, in the opinion of the Investigator or the Data Safety Monitoring Board compliance officer
  * postmenopausal female receiving HRT
  * pregnant or nursing
  * history of immunocompromise, including known HIV positivity as measured by enzyme-linked immunosorbent assay and western blot
  * active or suspected acute or chronic uncontrolled infection
  * history of noncompliance to medical regimens, potentially unreliability, or inability to complete the study
  * prior or concurrent radiotherapy for pituitary tumor
  * concurrent pituitary surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Heaney, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2006 - May 2009
Groups:
- Group 1 (ACTH-secreting Adenomas): Patients receive 4 mg oral rosiglitazone maleate once daily in week 1 and then 8 mg once daily beginning in week 2 and continuing for up to 6 months in the absence of disease progression or unacceptable toxicity.
  rosiglitazone maleate : Given orally
- Group 2 (Non-secreting Macroadenomas): Patients receive 4 mg oral rosiglitazone maleate once daily in week 1 and then 8 mg once daily beginning in week 2 and continuing for up to 12 months in the absence of disease progression or unacceptable toxicity.
  rosiglitazone maleate : Given orally
Period: Overall Study
Arm/Group | Group 1 (ACTH-secreting Adenomas) | Group 2 (Non-secreting Macroadenomas)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (ACTH-secreting Adenomas) | Group 2 (Non-secreting Macroadenomas) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Rosiglitazone Maleate on Cushing Disease
Description: Reduction in pituitary tumor volume by over 50% as assessed by MRI to measurements made at baseline.
Time Frame: 12 months
Population: No data was analyzed for this outcome measure as there was insufficient data to perform analysis.
Arm/Group | Group 1 (ACTH-secreting Adenomas) | Group 2 (Non-secreting Macroadenomas)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1 (ACTH-secreting Adenomas) | Group 2 (Non-secreting Macroadenomas)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Recruitment was the main limitation. Patients were available but were not interested in the study due to possible side effects of the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No